CLINICAL TRIAL: NCT04080440
Title: Stepped Wedge Cluster Randomised Controlled Trial to Assess the Readiness of Extubation in Brain-injured Patients Using a Clinical Score
Brief Title: Brain-injured Patients Extubation Readiness Study
Acronym: Biper
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: ANARLF Network (Unknown); Direction Générale de l'Offre de Soin (DGOS) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Biper - PhrcIR 2017 Chabanne; 2018-A00894-51 (Other: ANSM)
Record Dates: First submitted 2019-09-04; First posted 2019-09-06 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-02

CONDITIONS: Mechanical Ventilator Weaning; Acute Brain Injury; Altered Level of Consciousness; Mechanical Ventilation; Airway Control
Keywords: Coma; Intensive care units; Critical care; Stroke; Traumatic brain injury; Anoxic ischemic encephalopathy; Glasgow coma scale
MeSH Terms: conditions — Brain Injuries; Consciousness Disorders; Coma; Stroke; Brain Injuries, Traumatic; Hypoxia-Ischemia, Brain

STUDY DESIGN:
Intervention Model Description: Stepped wedge, cluster randomised controlled design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care (Active Comparator): Clinicians decide whether to extubate or not following usual care in their ICU ventilator weaning protocol
  Interventions: Procedure: Usual Care
- Extubation readiness clinical score (Experimental): Clinicians decide whether to extubate or not following the extubation readiness clinical score as part of their ICU ventilator weaning protocol
  Interventions: Procedure: Extubation readiness clinical score

INTERVENTIONS:
Procedure: Extubation readiness clinical score — After treatment of the acute neurological condition, eligibility for a spontaneous breathing trial will be assessed once a day.
  In the intervention group, after a successful spontaneous breathing trial in unconscious patients, the score will be evaluated.
  If the score is > 9, extubation has to be completed.
  Arms: Extubation readiness clinical score
Procedure: Usual Care — After treatment of the acute neurological condition, eligibility for a spontaneous breathing trial will be assessed once a day.
  In the control group, after a successful spontaneous breathing trial in unconscious patients, the extubation will be achieved according to usual care.
  Arms: Usual care

SUMMARY:
The BIPER study is a stepped wedge cluster randomised clinical trial aiming to decrease extubation failure in critically-ill brain-injured patients with residual impaired consciousness using a simple clinical score.

DETAILED DESCRIPTION:
Severe brain-injured patients need mechanical ventilation with tracheal intubation. After treatment of the acute neurological condition, weaning of the mechanical ventilation has to be initiated notably to prevent ventilator associated pneumonia and others complications. Nevertheless, extubation failure is very common in this population due to residual neurological impairment with airway control alteration.

Guidelines about weaning of mechanical ventilation and extubation exclude brain-injured patients with a residual impaired consciousness.

In 2017, a simple and pragmatic extubation readiness clinical score was validated in a prospective observational cohort study of 140 brain injured patients. (Godet et al. Anesthesiology. 2017 Jan;126(1):104-114) In this study, brain injured patients with residual impaired consciousness who succeeded a spontaneous breathing trial were extubated. In multivariate analysis, 4 clinical elements were associated with extubation success. A prediction score was determined using the odds ratio such as followed :

1. Deglutition: 3 points if present
2. Gag reflex: 4 points if present
3. Cough: 4 points if present
4. CRS-R Score, visual item >2, 3 points if present, 1 point if not

For a cut-off value of 9, extubation failure could be predicted with a sensibility of 84%, a specificity of 75%, a positive predictive value of 89% and a negative predictive value of 66%.

In order to participate, brain-injured patients will have to succeed a spontaneous breathing trial and meet all inclusion criteria, including not being able to obey to command with no or minimal sedation. Using a stepped wedge randomisation process with intensive care units as clusters, patients will be weaned and extubated under usual care or using the extubation readiness clinical score.

The authors' hypothesis is that this clinical score will allow physicians to extubate patients at the right time interval and prevent extubation failure in this frail population.

ELIGIBILITY:
Inclusion Criteria:

* Acute cerebral lesion with a Glasgow Coma Scale <13 needing admission in ICU and mechanical ventilation with tracheal intubation for neurological cause : cerebrovascular stroke either ischemic or hemorrhagic including aneurysmal subarachnoid hemorrhage, traumatic brain injury, anoxo ischemic encephalopathy after cardiac arrest or brain tumour
* Mechanical ventilation more than 48 hours
* 18 to 75 years old
* Neurological stability with no intracranial hypertension with minimal sedation
* Glasgow Coma Scale motor response < 6
* Spontaneous breathing trial succeeded
* First extubation attempt

Exclusion Criteria:

* Posterior cranial fossa lesion
* Admission for status epilepticus or central nervous system infection
* Spinal cord injury (tetraplegia or paraplegia)
* Uncontrolled status epilepticus or uncontrolled central nervous system infection
* Care limitation plan
* Chronic respiratory failure defined as ambulatory oxygen therapy or pressure support ventilation and/or proven COPD and/or ambulatory non-invasive CPAP therapy for sleep apnoea syndrome
* More than 3 failed spontaneous breathing trials
* Significant chest trauma (more than 2 broken ribs / broken sternum / with an indication of open thoracic surgery)
* Surgery planned within 7 days
* Tracheotomy or previous extubation outside of the protocol
* Previous compromised upper airway permeability
* Pregnant or breastfeeding woman
* Adult under the protection of the law or without social assurance system
* Inclusion in another clinical study about mechanical ventilation or weaning

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2020-02-09 (Actual); Primary Completion 2027-02-13 (Estimated); Study Completion 2027-10-13 (Estimated)

PRIMARY OUTCOMES:
Extubation failure | From extubation to Day 5 (120 hours) after extubation
  Extubation failure is defined as a need of reintubation or death in the 5 days (120 hours) following extubation

SECONDARY OUTCOMES:
Key secondary outcome measure: time to effective extubation | From enrollment to day 5 (120 hours) after extubation
  Time from SBT success (enrollment) to successful liberation from mechanical ventilation, defined as the time point at which a patient is alive and free of invasive ventilatory support for more than 5 days (120 hours)
Invasive mechanical ventilation duration | From admission to the end of ICU Stay
  Period expressed in days during which patients will need invasive mechanical ventilation
Non-invasive mechanical ventilation duration | From admission to the end of ICU Stay
  Period expressed in days during which patients will need non-invasive mechanical ventilation
Reintubation rate in the first 48 hours | From extubation to Day 2 after extubation (48 hours)
  Patients needing reintubation during the first 48h post-extubation
Reintubation rate in ICU | From extubation to the end of ICU Stay
  Patients needing reintubation during entire ICU stay
Post extubation nosocomial pneumonia | From extubation to the end of ICU stay
  Post extubation nosocomial pneumonia is defined as a pulmonary infection after extubation that necessitate antibiotic therapy
Tracheotomy after extubation | From extubation to the end of ICU Stay
  Number of patients that necessitate a tracheotomy after extubation failure
Tracheotomy before extubation | From enrollment to the end of ICU Stay
  Number of patients that necessitate a tracheotomy after a successful spontaneous breathing trial but before any extubation
ICU length of stay | From admission to the end of ICU Stay
  ICU length of stay expressed in days
Hospital length of stay | From admission to the end of Hospital Stay
  Hospital length of stay expressed in days
Mortality in ICU | From enrollment to the end of the ICU Stay
  Deceased patient in each group during ICU stay
Mortality at day 28 | From enrollment to Day 28
  Deceased patient in each group at day 28
Mortality at day 90 | From enrollment to Day 90
  Deceased patient in each group at day 90
Neurological outcome | Day 90 after enrollment
  Neurological outcome using the Glasgow Outcome Scale Extended

CONTACTS AND LOCATIONS:
Overall Officials: Russell Chabanne, Study Director — University Hospital, Clermont-Ferrand; Olivier Vincent, Principal Investigator — University Hospital, Grenoble; Florent Gobert, Principal Investigator — Hospices Civils de Lyon; Jérôme Morel, Principal Investigator — CHU SAINT-ETIENNE; Matthieu Jeannot, Principal Investigator — CH VALENCE; Pierre-André Rodié-Talbère, Principal Investigator — Nantes University Hospital; Thomas Geeraerts, Principal Investigator — University Hospital, Toulouse; Pierre-François Perrigault, Principal Investigator — University Hospital, Montpellier; Claire Roger, Principal Investigator — CHU Nîmes; Carole Ichai, Principal Investigator — CHU NICE; Nicolas Engrand, Principal Investigator — Fondation Ophtalmologique Adolphe de Rothschild; Camille Bouisse, Principal Investigator — CH de Bourg-en-Bresse; Natalie De Sa, Principal Investigator — CHU Lille; Sigismond Lasocki, Principal Investigator — University Hospital, Angers; Claire Dahyot-Fizelier, Principal Investigator — CHU Poitiers; Yoann Launey, Principal Investigator — CHU Rennes; Laurent Petit, Principal Investigator — CHU Bordeaux - Réanimation Chirurgicale et traumatologique; Hugues De Courson, Principal Investigator — CHU Bordeaux - Réanimation Neurologique; Clément Gakuba, Principal Investigator — CHU Caen Normandie; Sophie Kauffmann, Principal Investigator — CHU de La Réunion
Locations (20):
- France (20):
  - CHU, Angers
  - CHU, Bordeaux
  - CH, Bourg-en-Bresse
  - CHU, Caen
  - CHU, Clermont-Ferrand
  - CHU, Grenoble
  - CHU, La Réunion
  - CHU, Lille
  - Hospices Civils de Lyon, Lyon
  - APHM, Marseille
  - CHU, Montpellier
  - CHU, Nantes
  - Pasteur 2 Hospital - University Hospital, Nice
  - CHU, Nîmes
  - Fondation Ophtalmologique Adolphe de Rothschild, Paris
  - CHU, Poitiers
  - CHU, Rennes
  - CHU, Saint-Etienne
  - CHU, Toulouse
  - CH, Valence

IPD SHARING:
Plan to Share IPD: Yes
Data sharing plan : BIPER clinical trial data will be made available upon reasonable request as soon as study publication with deidentified participant data and statistical/analytic code
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: As soon as study publication in a peer review journal with a 5 years limit.
Access Criteria: Data will be made available on reasonable demand by emailing the coordinating clinical investigator of the trial. A proposal that describes planned analyses will have to be submitted and a data sharing agreement signed. Requests will be evaluated by the coordinating clinical investigator and study statistician of the trial.

REFERENCES:
- [Background] Godet T, Chabanne R, Marin J, Kauffmann S, Futier E, Pereira B, Constantin JM. Extubation Failure in Brain-injured Patients: Risk Factors and Development of a Prediction Score in a Preliminary Prospective Cohort Study. Anesthesiology. 2017 Jan;126(1):104-114. doi: 10.1097/ALN.0000000000001379. PMID 27749290
- [Derived] Chabanne R, Godet T, Andanson B, Borrel P, Astier L, Caumon E, Bourguignon N, Laclautre L, Morand D, De Jong A, Futier E, Constantin JM, Pereira B, Jabaudon M. Prevention of extubation failure in neurocritical care patients with residual disorder of consciousness: the Brain-Injured Patients Extubation Readiness (BIPER) study protocol for a stepped-wedge cluster-randomised controlled trial. BMJ Open. 2025 Jul 13;15(7):e104897. doi: 10.1136/bmjopen-2025-104897. PMID 40659406